CLINICAL TRIAL: NCT03605368
Title: Immersive Virtual Reality as a Tool to Improve Police Safety in Adolescents and Adults With ASD
Brief Title: VR Intervention to Improve Police Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Floreo, Inc. (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-014387; 1R42MH115539-01 (NIH)
Record Dates: First submitted 2018-07-23; First posted 2018-07-30 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Intervention; Technology
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase IIA - in-person (Active Comparator): Participants will be assigned to either a) a virtual reality-based intervention or b) an video modeling intervention both aimed at improving police interaction skills. Assessments of police skills will occur before intervention and after intervention (three sessions of each).
  Interventions: Behavioral: Virtual Reality Intervention; Behavioral: Video Modeling Intervention
- Phase IIB - remote (Active Comparator): Participants will be assigned to either a) three sessions of virtual reality-based intervention aimed at improving police interaction skills or b) no intervention. Assessments of police skills will occur before intervention, after intervention, and 3-4 weeks follow up in the intervention group and at comparable timepoints in the no intervention group.
  Interventions: Behavioral: Virtual Reality Intervention; Behavioral: No intervention

INTERVENTIONS:
Behavioral: Virtual Reality Intervention — Floreo's Police Safety Module (PSM) offers a supervised VR experience for people with ASD. The software is an application that provides a 3D immersive scene for headset-compatible smartphones. The person with ASD will use a smartphone capable of running the application with a dedicated headset providing the virtual environment. The PSM provides an immersive story-based intervention that shows a fully realized and intricately detailed urban environment designed to engage the user in a virtual encounter with a law enforcement officer. The immersive VR environment engages the person with ASD as an actor in a virtual narrative, incorporating strategies from both story-based intervention and video modeling. The video demonstrates the approach and initial engagement efforts of two police officers in the virtual environment, from the perspective of the person wearing the headset. The PSM allows a monitoring therapist to use a tablet or phone to supervise the person's virtual world.
Behavioral: Video Modeling Intervention — The video modeling intervention is a subset of the BE SAFE The Movie Curriculum Lessons (https://besafethemovie.com/curriculum/) that were selected to match Floreo PSM on length. The BE SAFE The Movie Curriculum consists of video-based instruction on police officer interaction expectations and safety. Within each of three sessions, participants will watch videos, complete worksheets, and discuss topics related to police safety knowledge and behaviors with the study administrator.
  Arms: Phase IIA - in-person
Behavioral: No intervention — Participants will follow all study procedures with the exception of the VR-based intervention including assessments.
  Arms: Phase IIB - remote

SUMMARY:
The primary objective of this study is to demonstrate the efficacy of Floreo's police safety module (PSM) in adolescents and adults with autism spectrum disorder (ASD) by assessing improvement in police interaction skills as compared to a video modeling intervention.

DETAILED DESCRIPTION:
Advances in virtual reality (VR) technology offer new opportunities to design interventions targeting the core deficits associated with autism spectrum disorder (ASD) and promote acquisition of skills necessary for effective navigation of challenging social situations, such as engagement with law enforcement. Researchers have explored the potential of virtual reality technology in targeting autism-related deficits, but at this time there are no evidence-based VR interventions for ASD. While most research labelled VR for the purposes of therapy has not been immersive, in recent years, the commercial introduction of head-mounted displays (HMD) and lower cost of virtual reality technology have led to greater interest in therapeutic applications of VR. As part of a mission to develop VR products for individuals with ASD, investigators will collaborate with a commercial tech start-up company, Floreo Technology, to study a mobile VR module for police safety skills. Investigators seek to evaluate the safety and feasibility of the mobile VR police safety module (PSM) and the effectiveness of the module in improving police interaction skills in adolescents and adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 12 to 60 years.
* Documented autism spectrum disorder (ASD) diagnosis
* Verbal Intelligence Quotient (IQ) >/= 75 (verbal and non-verbal)
* Informed consent (if adult) or parental/guardian permission (if child or adult with diminished capacity) and, if applicable, assent

Exclusion Criteria:

* Participation in pilot virtual reality (VR) study at the Children's Hospital of Philadelphia (CHOP)
* Personal or family history of seizures or a seizure disorder
* Primary sensory impairment (e.g., blindness, deafness)
* Personal or family history of migraines
* History of vertigo
* History of strabismus, other eye muscle problems, or eye surgery
* History of concussion with hospitalization
* Diagnosis of a known genetic syndrome (e.g., Down syndrome, Fragile X syndrome)
* History of a medical condition which has affected/affects cognitive, sensory, or motor functioning (e.g., Fetal Alcohol Syndrome, brain injury, stroke, brain tumor)
* Non-English speaking
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 158 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Parish-Morris, PhD, Principal Investigator — Children's Hospital of Philadelphia; Vijay Ravindran, Principal Investigator — Floreo, Inc.
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 158 individuals enrolled, 28 did not meet inclusion criteria (low IQ scores), and we could not confirm eligibility for 18 individuals due to lost contact.
Groups:
- Phase IIA - In-Person Floreo PSM; Phase IIA - In-Person BeSAFE Video Modeling: Participants will be assigned to either (a) a virtual reality-based intervention or (b) a video modeling intervention, both aimed at improving police interaction skills. Assessments of police interaction skills will occur in-person before/after intervention (three sessions of each, separated by approximately 1 week).
  Virtual Reality Intervention: Floreo's Police Safety Module (PSM) is a 3D immersive story-based intervention designed to engage the user in a virtual encounter with a law enforcement officer. The immersive VR environment engages the person as an actor in a virtual narrative, incorporating strategies from both story-based intervention and video modeling to practice social skills. The video demonstrates the approach and initial engagement efforts of two police officers in the virtual environment, from the perspective of the person wearing the headset. The PSM allows a monitoring therapist to use a tablet or phone to supervise the person's virtual world.
  Video Modeling Intervention: The video modeling intervention is a subset of the BE SAFE The Movie Curriculum Lessons (https://besafethemovie.com/curriculum/) that were selected to match Floreo PSM on length. The BE SAFE The Movie Curriculum consists of video-based instruction on police officer interaction expectations and safety. Within each of three sessions, participants will watch videos, complete worksheets, and discuss topics related to police safety knowledge and behaviors with the study administrator.
- Phase IIB - Remote Floreo PSM; Phase IIB - Remote Treatment-As-Usual (TAU): Participants will be assigned to either (a) three sessions of remote at-home virtual reality-based intervention aimed at improving police interaction skills or (b) no intervention (treatment-as-usual, TAU). Remote videoconference-based assessments of police skills will occur before intervention, after intervention, and 3-4 weeks follow-up in the intervention group and at comparable timepoints in the no intervention group.
  Virtual Reality Intervention: Floreo's Police Safety Module (PSM) is a 3D immersive story-based intervention designed to engage the user in a virtual encounter with a law enforcement officer. The immersive VR environment engages the person as an actor in a virtual narrative, incorporating strategies from both story-based intervention and video modeling to practice social skills. The video demonstrates the approach and initial engagement efforts of two police officers in the virtual environment, from the perspective of the person wearing the headset. The PSM allows a monitoring therapist to use a tablet or phone to supervise the person's virtual world via videoconference.
  No intervention: Participants will follow all study procedures with the exception of the VR-based intervention including assessments.
Period: Overall Study
Arm/Group | Phase IIA - In-Person Floreo PSM | Phase IIA - In-Person BeSAFE Video Modeling | Phase IIB - Remote Floreo PSM | Phase IIB - Remote Treatment-As-Usual (TAU)
Started | 25 | 25 | 31 | 31
Completed | 23 | 24 | 24 | 26
Not Completed | 2 | 1 | 7 | 5
Not completed — Lost to Follow-up | 2 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Population: Baseline participants is taken to mean participants that completed the study and included in the final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase IIA - In-Person Floreo PSM | Phase IIA - In-Person BeSAFE Video Modeling | Phase IIB - Remote Floreo PSM | Phase IIB - Remote Treatment-As-Usual (TAU) | Total
Number analyzed (Participants) | 23 | 24 | 24 | 26 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two participants in Phase IIB have missing age information: 1 Floreo PSM, 1 TAU.
  years
    number analyzed (Participants) | 23 | 24 | 23 | 25 | 95
    (all) | 21.87 (10.50) | 21.50 (11.44) | 18.26 (6.29) | 19.92 (8.39) | 20.39 (9.16)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex assigned at birth: Female | 4 | 4 | 10 | 11 | 29
  Sex assigned at birth: Male | 19 | 20 | 14 | 15 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 4 | 2 | 9
  Not Hispanic or Latino | 21 | 23 | 20 | 24 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 5 | 1 | 14
  White | 14 | 20 | 16 | 22 | 72
  More than one race | 2 | 1 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 24 | 26 | 97
Wechsler Abbreviated Scale of Intelligence - 2nd Edition [Mean (Standard Deviation); unit: units on a scale] — The Wechsler Abbreviated Scale of Intelligence - Second Edition is a measure designed to estimate full-scale intelligence quotient (FSIQ). The FSIQ provides an overall estimate of an individual's general intellectual ability, with a mean of 100 and a standard deviation of 15 (range: 40-160). Higher scores indicate greater estimated intellectual ability. Population: In Phase IIB, two participants had missing IQ information (1 Floreo PSM, 1 TAU).
  units on a scale
    number analyzed (Participants) | 23 | 24 | 23 | 25 | 95
    (all) | 100.70 (15.52) | 102.92 (14.36) | 102.26 (14.60) | 104.00 (13.15) | 102.47 (14.41)
Autism Diagnosis [Count of Participants; unit: Participants] | 23 | 24 | 24 | 26 | 97

OUTCOME MEASURES:

1. Primary Outcome: Change in Live or Virtual Police Interaction Assessment Scores From Pre-to-Post Treatment
Description: The primary efficacy endpoint is the change in live in-person (Phase IIA) or virtual (Phase IIB) Police Interaction Assessment Scores between the Floreo PSM Virtual Reality Intervention and BE SAFE Video-Based intervention (Phase IIA) or treatment-as-usual (Phase IIB) from pre-treatment to post-treatment. Greater pre-treatment to post-treatment scores indicate better 3rd party ratings of social skills in that domain. The range of possible scores for the Police Interaction Assessment is -3 (performance got significantly worse from pre-treatment to post-treatment) to 3 (performance improved significantly from pre-treatment to post-treatment) on each variable (overall behavior, appropriate response, orienting, and fidgeting).
Time Frame: The Police Interaction Assessment was administered pre- and post-intervention (~2 weeks apart). Outcome measure data represent the difference in Police Interaction Assessment scores (post-intervention minus pre-intervention.)
Population: The analysis population is described in Baseline Characteristics.
Measure: Mean (Standard Deviation); unit: Change from baseline - units on a scale
Arm/Group | Phase IIA - In-Person Floreo PSM | Phase IIA - In-Person BeSAFE Video Modeling | Phase IIB - Remote Floreo PSM | Phase IIB - Remote Treatment-As-Usual (TAU)
Number analyzed (Participants) | 23 | 24 | 24 | 26
Change from baseline - units on a scale
  Overall Behavior | .13 (.42) | .29 (.50) | -.28 (.39) | .02 (.41)
  Appropriate Response | .04 (.29) | .21 (.35) | -.13 (.34) | .06 (.29)
  Orienting | .18 (.49) | .18 (.66) | -.14 (.46) | .20 (.73)
  Fidgeting | -.03 (.56) | .44 (.52) | -.31 (.53) | -.07 (.45)
Statistical Analysis 1: Comparison: Phase IIA - In-Person Floreo PSM vs Phase IIA - In-Person BeSAFE Video Modeling; Overall Behavior. Change-from-baseline analyses were conducted (post-intervention assessment ratings minus pre-intervention assessment ratings) and compared between intervention groups (Floreo and BeSAFE); Test type: Equivalence — Simple linear models ('lm' in R) were conducted. Statistical significance was set at p<.05; p = .23, Regression, Linear; Mean Difference (Final Values) = .16, Standard Error of Mean .13
Statistical Analysis 2: Comparison: Phase IIA - In-Person Floreo PSM vs Phase IIA - In-Person BeSAFE Video Modeling; Appropriate Response. Change-from-baseline analyses were conducted (post-intervention assessment ratings minus pre-intervention assessment ratings) and compared between intervention groups (Floreo and BeSAFE); Test type: Equivalence — Simple linear models ('lm' in R) were conducted. Statistical significance was set at p<.05; p = .07, Regression, Linear; Mean Difference (Final Values) = .17, Standard Error of Mean .09
Statistical Analysis 3: Comparison: Phase IIA - In-Person Floreo PSM vs Phase IIA - In-Person BeSAFE Video Modeling; Orienting. Change-from-baseline analyses were conducted (post-intervention assessment ratings minus pre-intervention assessment ratings) and compared between intervention groups (Floreo and BeSAFE); Test type: Equivalence — Simple linear models ('lm' in R) were conducted. Statistical significance was set at p<.05; p = .99, Regression, Linear; Mean Difference (Final Values) = -.00, Standard Error of Mean .17
Statistical Analysis 4: Comparison: Phase IIA - In-Person Floreo PSM vs Phase IIA - In-Person BeSAFE Video Modeling; Fidget. Change-from-baseline analyses were conducted (post-intervention assessment ratings minus pre-intervention assessment ratings) and compared between intervention groups (Floreo and BeSAFE); Test type: Equivalence — Simple linear models ('lm' in R) were conducted. Statistical significance was set at p<.05; p = .005, Regression, Linear; Mean Difference (Final Values) = .47, Standard Error of Mean .16
Statistical Analysis 5: Comparison: Phase IIB - Remote Floreo PSM vs Phase IIB - Remote Treatment-As-Usual (TAU); Overall Behavior. Change-from-baseline analyses were conducted (post-intervention assessment ratings minus pre-intervention assessment ratings) and compared between intervention groups (Floreo and TAU); Test type: Equivalence — Simple linear models ('lm' in R) were conducted. Statistical significance was set at p<.05; p = .01, Regression, Linear; Mean Difference (Final Values) = .30, Standard Error of Mean .11
Statistical Analysis 6: Comparison: Phase IIB - Remote Floreo PSM vs Phase IIB - Remote Treatment-As-Usual (TAU); Appropriate Response. Change-from-baseline analyses were conducted (post-intervention assessment ratings minus pre-intervention assessment ratings) and compared between intervention groups (Floreo and TAU); Test type: Equivalence — Simple linear models ('lm' in R) were conducted. Statistical significance was set at p<.05; p = .04, Regression, Linear; Mean Difference (Final Values) = .19, Standard Error of Mean .09
Statistical Analysis 7: Comparison: Phase IIB - Remote Floreo PSM vs Phase IIB - Remote Treatment-As-Usual (TAU); [analysis description as in outcome 1, analysis 6]; Test type: Equivalence — Simple linear models ('lm' in R) were conducted. Statistical significance was set at p<.05; p = .06, Regression, Linear; Mean Difference (Final Values) = .34, Standard Error of Mean .17
Statistical Analysis 8: Comparison: Phase IIB - Remote Floreo PSM vs Phase IIB - Remote Treatment-As-Usual (TAU); Test type: Equivalence — Simple linear models ('lm' in R) were conducted. Statistical significance was set at p<.05; p = .09, Regression, Linear; Mean Difference (Final Values) = .24, Standard Error of Mean .14

2. Secondary Outcome: Change in Police Interaction Knowledge
Description: The secondary endpoint includes changes in Police Interaction Knowledge Questionnaire Scores from Pre-Treatment to Post-Treatment or Pre-TAU to Post-TAU. Before and after the in-person Floreo VR intervention, participants completed a 10-question survey that asked about their feelings of comfort and safety when interacting with police officers. The scale for each question ranged from 1-7, with 7 indicating greater feelings of safety, comfort, and knowledge and 1 indicating fewer feelings of safety, comfort, and knowledge. Scores were summed to create a total score, which ranged from 10 to 70, and then subtracted to calculate a change score (post-intervention minus pre-intervention). Change scores, which had a possible range of -60 to +60, were compared between groups. Greater change scores after intervention or TAU indicate greater feelings of safety, comfort, and knowledge when interacting with police.
Time Frame: Baseline and immediately post-intervention (~2 weeks apart)
Population: The analysis population is described in Baseline Characteristics. Missing data: In Phase IIA, no data are missing. In Phase IIB, 6 participants in the Floreo condition and 3 in the TAU condition are missing Police Interaction Knowledge questionnaire data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase IIA - In-Person Floreo PSM | Phase IIA - In-Person BeSAFE Video Modeling | Phase IIB - Remote Floreo PSM | Phase IIB - Remote Treatment-As-Usual (TAU)
Number analyzed (Participants) | 23 | 24 | 18 | 23
units on a scale | 8.09 (9.54) | 9.71 (8.68) | 8.11 (9.09) | 2.70 (8.35)
Statistical Analysis 1: Comparison: Phase IIA - In-Person Floreo PSM vs Phase IIA - In-Person BeSAFE Video Modeling; Test type: Equivalence — A linear regression compared change in Police Interaction Knowledge scores by group (Floreo vs. TAU) from pre- to post-intervention. Significance was set at p<.05; p = .55, Regression, Linear; Mean Difference (Final Values) = 1.62, Standard Error of Mean 2.67
Statistical Analysis 2: Comparison: Phase IIB - Remote Floreo PSM vs Phase IIB - Remote Treatment-As-Usual (TAU); Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = .05, Regression, Linear; Mean Difference (Final Values) = 5.42, Standard Error of Mean 2.73

ADVERSE EVENTS:
Time Frame: Adverse events were monitored by study staff at baseline, during intervention or TAU, at the post-intervention assessment, and at follow-up. Monitoring continued through study completion, which was an average of 2 weeks for Phase IIA and 6 weeks for Phase IIB.
Description: No series adverse events occurred.
Groups:
- Phase IIA - In-person: Participants will be assigned to either (a) a virtual reality-based intervention or (b) a video modeling intervention, both aimed at improving police interaction skills. Assessments of police interaction skills will occur in-person before/after intervention (three sessions of each, separated by approximately 1 week).
  Virtual Reality Intervention: Floreo's Police Safety Module (PSM) is a 3D immersive story-based intervention designed to engage the user in a virtual encounter with a law enforcement officer. The immersive VR environment engages the person as an actor in a virtual narrative, incorporating strategies from both story-based intervention and video modeling to practice social skills. The video demonstrates the approach and initial engagement efforts of two police officers in the virtual environment, from the perspective of the person wearing the headset. The PSM allows a monitoring therapist to use a tablet or phone to supervise the person's virtual world.
  Video Modeling Intervention: The video modeling intervention is a subset of the BE SAFE The Movie Curriculum Lessons (https://besafethemovie.com/curriculum/) that were selected to match Floreo PSM on length. The BE SAFE The Movie Curriculum consists of video-based instruction on police officer interaction expectations and safety. Within each of three sessions, participants will watch videos, complete worksheets, and discuss topics related to police safety knowledge and behaviors with the study administrator.
- Phase IIB - Remote: Participants will be assigned to either (a) three sessions of remote at-home virtual reality-based intervention aimed at improving police interaction skills or (b) no intervention (treatment-as-usual, TAU). Remote videoconference-based assessments of police skills will occur before intervention, after intervention, and 3-4 weeks follow-up in the intervention group and at comparable timepoints in the no intervention group.
  Virtual Reality Intervention: Floreo's Police Safety Module (PSM) is a 3D immersive story-based intervention designed to engage the user in a virtual encounter with a law enforcement officer. The immersive VR environment engages the person as an actor in a virtual narrative, incorporating strategies from both story-based intervention and video modeling to practice social skills. The video demonstrates the approach and initial engagement efforts of two police officers in the virtual environment, from the perspective of the person wearing the headset. The PSM allows a monitoring therapist to use a tablet or phone to supervise the person's virtual world via videoconference.
  No intervention: Participants will follow all study procedures with the exception of the VR-based intervention including assessments.
Arm/Group | Phase IIA - In-person | Phase IIB - Remote
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/50
Other Adverse Events (participants affected / at risk) | 0/47 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT03605368/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03605368/ICF_001.pdf